CLINICAL TRIAL: NCT03280706
Title: Gastric Emptying of Maltodextrin Compared to Coffee With Milk and Orange Juice During Labor at Term: Non-inferiority Clinical Trial
Brief Title: Gastric Emptying During Labor at Term: Non-inferiority Clinical Trial
Acronym: GEMCO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brasilia University Hospital (Other)
Responsible Party: Principal Investigator, Gabriel Magalhaes Nunes Guimaraes, Head of anesthesiology, Brasilia University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: tcc-anele-2017
Record Dates: First submitted 2017-09-09; First posted 2017-09-12 (Actual); Last update posted 2018-02-07 (Actual); Status verified 2018-02

CONDITIONS: Gastric Emptying; Pregnancy Vomits
Keywords: Gastric Emptying; labor; maltodextrin; orange juice; coffee; ultrasound
MeSH Terms: interventions — maltodextrin; Coffee; Milk

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Investigator and outcomes assessor will not know to which group each woman was allocated
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Maltodextrin (Experimental): Fasted pregnant woman with an empty stomach (assessed by ultrasound) will drink 500ml of maltodextrin 200kcal, no protein or fat, 49,5g of carbohydrate.
  Interventions: Dietary Supplement: Maltodextrin
- Orange Juice (Active Comparator): Fasted pregnant woman with an empty stomach (assessed by ultrasound) will drink 500ml of orange juice, 200kcal, 2,82g of protein, 0,67g of fat, 47,08g of carbohydrate.
  Interventions: Dietary Supplement: Orange Juice
- Coffee with milk (Active Comparator): Fasted pregnant woman with an empty stomach (assessed by ultrasound) will drink 500ml of coffee with milk, 200kcal, 10,6g of protein, 10,73g of fat, 14,9g of carbohydrate.
  Interventions: Dietary Supplement: Coffee with milk

INTERVENTIONS:
Dietary Supplement: Maltodextrin — Maltodextrin 50g in water 500ml
  Arms: Maltodextrin
Dietary Supplement: Orange Juice — Orange juice 480ml + 20ml of water
  Arms: Orange Juice
Dietary Supplement: Coffee with milk — Coffee with milk (330 ml of milk + 220 of water)
  Arms: Coffee with milk

SUMMARY:
This study evaluates the gastric emptying of pregnant woman at term who received one of the three solutions: maltodextrin, orange juice or coffee with milk.

DETAILED DESCRIPTION:
Allocation in maltodextrin, orange juice or coffee with milk will be random using sealed envelopes. Gastric ultrasound will be used for estimating gastric volume by measuring antral area in right lateral decubiti. All solutions will have the same volume and total of calories.

ELIGIBILITY:
Inclusion Criteria:

* Pregnancy at term
* Fasted with an emptying stomach (assessed by ultrasound)
* During Labor
* No diabetes, esophageal disease, obesity
* Not emergency
* High risk of need of general anesthesia

Exclusion Criteria:

* Vomiting before the end of the protocol
* Did not drink the whole solutions
* Ultrasound not performed for any reason

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2017-09-09 (Actual); Primary Completion 2018-02-01 (Actual); Study Completion 2018-02-02 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Gastric antral area | baseline (before drinking allocated solution), 30, 60, 90 and 120 minutes after drinking.
  Change from Baseline Gastric antral area measured by ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel MN Guimaraes, MsC, Study Chair — Hospital Universitario de Brasilia
Locations (1):
- University Hospital of Brasilia University, Brasília, Federal District, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Will make it available in our website
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 6 months after the end of the study
Access Criteria: Open access
URL: http://www.anestesiologiaunb.com.br